CLINICAL TRIAL: NCT07103850
Title: Suicidal Crisis Syndrome and the Suicide Crisis Inventory-Revised (SCS-2): Psychometric Properties of the Spanish Version
Brief Title: Latin American Testing of the Inventory for Risk in Suicidal Crisis Syndrome (LATIR-SCS)
Acronym: LATIR-SCS
Status: Recruiting | Type: Observational
Sponsor: University Diego Portales (Other)
Collaborators: Hospital Dr Sotero del Rio (Other)
Responsible Party: Principal Investigator, Francisco Javier Villalon Lopez, Principal Investigator, University Diego Portales
Other Study IDs: 071124
Record Dates: First submitted 2025-07-21; First posted 2025-08-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Suicidal Crisis
Keywords: Suicidal Crisis Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCS+ Cohort: Definition: Patients who meet the diagnostic criteria for Suicidal Crisis Syndrome using the clinician-administered SCS-C.
  Interventions: Diagnostic Test: Suicidal Crisis Syndrome Checklist (SCS-C); Diagnostic Test: Suicide Crisis Inventory-Revised (SCS-2)
- SCS- Cohort: Definition: Patients hospitalized for suicidal behavior who do not meet diagnostic criteria for SCS on the SCS-C.
  Interventions: Diagnostic Test: Suicidal Crisis Syndrome Checklist (SCS-C); Diagnostic Test: Suicide Crisis Inventory-Revised (SCS-2)

INTERVENTIONS:
Diagnostic Test: Suicidal Crisis Syndrome Checklist (SCS-C) — The Suicidal Crisis Syndrome Checklist (SCS-C) is a clinician-rated tool designed to diagnose Suicidal Crisis Syndrome (SCS), a suicide-specific state associated with imminent risk. It includes Criterion A (entrapment)-a required symptom-and Criterion B, which requires at least one symptom from each of four domains: affective disturbance, loss of cognitive control, hyperarousal, and social withdrawal. The checklist offers a structured assessment for identifying acute suicide risk, complementing traditional risk evaluations.
Diagnostic Test: Suicide Crisis Inventory-Revised (SCS-2) — The Suicide Crisis Inventory-Revised (SCS-2) is a 61-item self-report scale developed to assess the severity of Suicidal Crisis Syndrome (SCS), a clinical state associated with imminent suicide risk. Items are rated on a Likert scale and grouped into five empirically derived factors: entrapment, affective disturbance, loss of cognitive control, hyperarousal, and social withdrawal. The SCS-2 has shown strong internal consistency and predictive validity for suicidal behavior within weeks of discharge. It is currently undergoing cultural adaptation and psychometric validation in Spanish for use in high-risk psychiatric populations in Chile.

SUMMARY:
The goal of this observational validation study is to assess the psychometric properties of the Spanish versions of the Suicide Crisis Inventory-Revised (SCS-2) and the Suicidal Crisis Syndrome Checklist (SCS-C) in adults recently hospitalized for suicidal behavior in Chile. The study aims to determine whether the Spanish versions of the SCS-2 and SCS-C demonstrate adequate internal consistency, construct validity, interrater reliability, and test-retest stability, and whether these tools validly assess imminent suicide risk in a Spanish-speaking psychiatric population. Clinical assessments using the SCS-2 and SCS-C will be compared with established diagnostic and functional measures, including the Mini International Neuropsychiatric Interview (MINI), the Sheehan Disability Scale (SDS), and the Sheehan Suicidality Tracking Scale (S-STS), to evaluate convergent and discriminant validity. Participants will complete the SCS-2 and SCS-C at both admission and discharge from a psychiatric intensive care unit, undergo structured interviews and functional assessments, be evaluated by two independent raters for interrater reliability, and be reassessed within a short time interval to measure test-retest reliability. Follow-up contacts at 7 and 30 days post-discharge will be used to assess suicidal behavior outcomes. This is the first study to culturally adapt and validate these suicide-specific instruments in Latin America.

DETAILED DESCRIPTION:
This is a three-phase, observational psychometric validation study of the Spanish versions of the Suicide Crisis Inventory-Revised (SCS-2) and the Suicidal Crisis Syndrome Checklist (SCS-C), administered to adult psychiatric inpatients hospitalized for recent suicidal behavior at the Complejo Asistencial Dr. Sótero del Río (CASR), Chile. The study follows established guidelines for the translation, cultural adaptation, and validation of health-related instruments. Phase one involves linguistic validation through forward-backward translation by bilingual experts. Phase two consists of a pilot test of the pre-final versions with 10 patients to assess item clarity and cultural relevance. Phase three uses a prospective cohort design with 60 participants to evaluate psychometric properties. Assessments are conducted at admission and discharge and include the SCS-2 and SCS-C (Spanish versions), the Mini International Neuropsychiatric Interview (MINI), the Sheehan Disability Scale (SDS), and the Sheehan Suicidality Tracking Scale (S-STS). A subset of participants will complete the SCS-2 twice within a short time interval to assess test-retest reliability and will be evaluated by two independent raters for interrater reliability. Follow-up at 7 and 30 days post-discharge includes phone interviews and chart reviews to assess suicidal behavior outcomes. A sample size of 60 was selected based on prior studies to ensure sufficient power to evaluate internal consistency (Cronbach's α ≥ 0.80), factor structure, and interrater reliability (Cohen's κ ≥ 0.60). Statistical analyses will include Cronbach's alpha and item-total correlations for internal consistency, exploratory and confirmatory factor analysis (EFA/CFA) for construct validity, Pearson or Spearman correlations with SDS and S-STS for convergent validity, point-biserial correlations with MINI diagnoses for discriminant validity, ICC and Cohen's kappa for interrater reliability, ICC for test-retest reliability, and ROC curve analysis for predictive validity. Data will be collected electronically via Qualtrics, which includes built-in logic checks and skip patterns. Source data verification will be performed through cross-checks with clinical records and dual entry of outcome events. A detailed data dictionary outlines all variables, coding schemes, and response formats. Procedures are standardized through SOPs covering recruitment, consent, data collection, follow-up, and confidentiality. Missing data will be addressed through multiple imputation and sensitivity analyses. Data monitoring is performed internally, and adverse events or protocol deviations are reported to the Institutional Ethics Committee. This is the first study to validate the SCS-2 and SCS-C in a Spanish-speaking Latin American population and is expected to contribute to scalable, evidence-based suicide risk assessments in acute psychiatric settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Currently hospitalized in the Psychiatric Intensive Care Unit (UHCIP) at Complejo Asistencial Dr. Sótero del Río (CASR)
* Hospitalization due to a recent suicidal event, defined as at least one of the following:

  1. Deliberate self-inflicted violence with actual or potential injury and explicit or implicit suicidal intent
  2. Preparatory behaviors for suicide
  3. Aborted suicide attempts
  4. Interrupted suicide attempts
  5. Suicidal ideation leading to emergency consultation or referral
* Able to provide informed consent
* Judged competent to participate by the treating psychiatrist
* Fluent in Spanish

Exclusion Criteria:

* Presence of severe psychotic symptoms
* Qualitative or quantitative disturbance of consciousness (e.g., delirium, coma)
* Severe psychomotor agitation requiring mechanical restraint
* Inability to understand or complete study procedures (e.g., due to cognitive impairment or language barriers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult psychiatric inpatients (≥18 years old) hospitalized in the Psychiatric Intensive Care Unit (UHCIP) of the Complejo Asistencial Dr. Sótero del Río (CASR), Santiago, Chile. All participants are admitted due to a recent suicidal event, including suicide attempts, preparatory behaviors, interrupted or aborted attempts, or suicidal ideation requiring emergency care. The sample includes individuals with diverse psychiatric diagnoses and varying levels of acute suicide risk. Participants must be clinically stable, capable of providing informed consent, and fluent in Spanish. The population is representative of high-risk individuals typically seen in public psychiatric emergency settings in Latin America.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal Event Within 30 Days Post-Discharge | 30 days post-discharge
  Description: Occurrence of a suicidal event within 30 days after discharge, defined as any of the following:
  1. Deliberate self-inflicted violence resulting in actual or potential injury, with explicit or implicit evidence of suicidal intent;
  2. Preparatory behaviors for suicide;
  3. Aborted suicide attempts;
  4. Interrupted suicide attempts; or
  5. Suicidal ideation leading to emergency consultation or referral.
  Assessment Method: Patient phone follow-up and review of clinical records Measure Type: Clinical outcome (binary: presence/absence of suicidal event)

SECONDARY OUTCOMES:
Suicidal Event Within 7 Days Post-Discharge | 7 days post-discharge
  Description: Occurrence of a suicidal event within 7 days after discharge, defined as any of the following:
  1. Deliberate self-inflicted violence resulting in actual or potential injury, with explicit or implicit evidence of suicidal intent;
  2. Preparatory behaviors for suicide;
  3. Aborted suicide attempts;
  4. Interrupted suicide attempts; or
  5. Suicidal ideation leading to emergency consultation or referral.
  Assessment Method: Patient phone follow-up and review of clinical records Measure Type: Clinical outcome (binary: presence/absence of suicidal event)
Convergent Validity with the Sheehan Suicidality Tracking Scale (S-STS) | Baseline
  Description: Strength of association between total scores on the Spanish SCS-2, SCS-C and S-STS, a validated measure of suicidal risk severity.
  Assessment Method: Pearson or Spearman correlation coefficients Measure Type: Psychometric validity (convergent)
Convergent Validity with the Sheehan Disability Scale (SDS) | Baseline
  Description: Correlation between SCS-2 total scores, SCS-C and functional impairment measured by the SDS in three domains: work, social life, and family responsibilities.
  Assessment Method: Pearson or Spearman correlations Measure Type: Psychometric validity (convergent)
Discriminant Validity with Psychiatric Diagnoses on the MINI | Baseline
  Description: Ability of the SCS-2 and SCS-C to discriminate between participants with and without current psychiatric diagnoses commonly associated with elevated suicide risk, as assessed by the Mini International Neuropsychiatric Interview (MINI). Diagnoses of interest include:
  Major Depressive Episode Post-Traumatic Stress Disorder (PTSD) Panic Disorder
  Assessment Method: Point-biserial correlations and group comparisons Measure Type: Psychometric validity (discriminant)
Test-Retest Reliability of the SCS-2 | Up to 48 hours from baseline
  Description: Stability of SCS-2 scores across two administrations within a short interval (24-48 hours) during hospitalization, in the absence of clinical change.
  Assessment Method: Intraclass correlation coefficient (ICC) Measure Type: Reliability (test-retest)
Interrater Reliability of the SCS-C (Spanish version) | Up to 48 hours from baseline
  Description: Agreement between two independent raters administering the SCS-C to the same participant within the same time frame.
  Assessment Method: Intraclass correlation coefficient (ICC) and Cohen's kappa Measure Type: Reliability (interrater)
Internal Consistency of the SCS-2 (Spanish Version) | Baseline
  Description: Evaluation of the psychometric properties of the Spanish version of the SCS-2, including internal consistency (Cronbach's alpha and item-total correlations). The goal is to assess the reliability of the total scale.
  Assessment Method: Cronbach's alpha, item-total correlations Measure Type: Reliability (internal consistency)
Internal Consistency of the SCS-C (Spanish Version) | Baseline
  Description: Evaluation of the psychometric properties of the Spanish version of the SCS-C, including internal consistency (Kuder-Richardson 20). The goal is to assess the reliability of the total scale.
  Assessment Method: Kuder-Richardson 20 Measure Type: Reliability (internal consistency)
Construct Validity of the SCS-2 (Spanish Version) | Baseline
  Description: Evaluation of the psychometric properties of the Spanish version of the SCS-2, including construct validity through exploratory and confirmatory factor analyses. The goal is to confirm the five-factor structure: entrapment, affective disturbance, cognitive dyscontrol, hyperarousal, and social withdrawal.
  Assessment Method: Exploratory Factorial Analysis, and Confrimatory Factorial Analysis with fit indices (e.g., CFI, TLI, RMSEA, SRMR) Measure Type: Psychometric validity (construct validity)
Construct Validity of the SCS-C (Spanish Version) | Baseline
  Description: Evaluation of the psychometric properties of the Spanish version of the SCS-C, including construct validity through exploratory and confirmatory factor analyses. The goal is to confirm the five-factor structure: entrapment, affective disturbance, cognitive dyscontrol, hyperarousal, and social withdrawal.
  Assessment Method: Exploratory Factorial Analysis, and Confrimatory Factorial Analysis with fit indices (e.g., CFI, TLI, RMSEA, SRMR) Measure Type: Psychometric validity (construct validity)
Concurrent Validity of the SCS-2 and SCS-C (Spanish Versions) | Baseline
  Description: Evaluation of the psychometric properties of the Spanish versions of the SCS-2 and SCS-C, including concurrent validity through the correlation of their total and subscale scores when administered at the same time. The primary goal is to verify whether the two formats (Likert and dichotomous checklist) consistently measure the construct of suicidal crisis syndrome. Correlations will be calculated using Pearson or Spearman coefficients for total and subscale scores. Additionally, point-biserial correlations will be conducted at the item level to further examine the association between dichotomous responses on the SCS-C and continuous scores on the corresponding dimensions of the SCS-2.
  Assessment Method: Pearson/Spearman correlations for total and subscale scores; point-biserial correlations for item-level analysis.
  Measure Type: Psychometric validity (concurrent). Time Frame: Baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Asistencial Sotero del Rio, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
e-identified individual participant data (IPD) underlying the published results may be shared upon reasonable request and prior approval by the institutional Ethics Committee. Data sharing will be considered for academic, non-commercial purposes only, and requires submission of a data use proposal outlining objectives, analysis plan, and measures for confidentiality protection.